CLINICAL TRIAL: NCT05673824
Title: Effect of Huaier Granule on Nephrotoxicity Associated With Anti-angiogenesis Targeted Therapy for Advanced Hepatobiliary Malignancies: a Single-arm, Single-center, Exploratory Study.
Brief Title: Effect of Huaier Granule on Nephrotoxicity Associated With Targeted Therapy for Advanced Hepatobiliary Malignancies.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: LinkDoc Technology (Beijing) Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Lu Wang, MD, PhD, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE-202210
Record Dates: First submitted 2022-12-21; First posted 2023-01-06 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Nephrotoxicity
Keywords: Huaier granule; proteinuria; hepatobiliary malignancies; anti-angiogenesis targeted therapy
MeSH Terms: conditions — Proteinuria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Huaier Granule Group (Experimental): Huaier Granule+VEGFR-TKIs
  Interventions: Drug: Huaier Granule; Drug: VEGFR-TKIs

INTERVENTIONS:
Drug: Huaier Granule — Treatment period: oral administration, 10g each time, 3 times a day. Continuous medication until the end of the study, failure of treatment, intolerable toxicity, withdrawal from the study for any reason or death, whichever occurs first; or after researcher's judgement, patient would no longer benefit from the treatment.
  If the treatment of hepatobiliary malignancies needs to be changed due to disease progression, whether to continue the medication or not should be determined by the researcher.
Drug: VEGFR-TKIs — Treatment period: Therapeutic agents were selected according to clinical routine, including but not limited to Sorafenib, Lenvatinib, Donafenib, Regorafenib, Apatinib and Cabozantinib. Continuous medication until disease progression, intolerable toxicity, withdrawal from the study for any reason or death, whichever occurs first. Refer to drug instructions for specific usage.

SUMMARY:
This is a prospective, single-arm, single-center, exploratory study. The purpose of this study is to explore the effect of Huaier Granule on nephrotoxicity associated with anti-angiogenesis targeted therapy for advanced hepatobiliary malignancies.

DETAILED DESCRIPTION:
China is a country with a high incidence of liver cancer, and the incidence of primary liver cancer ranks the fourth among malignant tumors in China. Hepatocellular carcinoma (HCC) is the main type of liver cancer, accounting for 75% to 85%. About 39.0%-53.6% of HCC patients were already advanced when first visit and had lost the opportunity to receive radical treatment. Currently, anti-angiogenesis targeted drugs are recommended for the first- or second-line treatment of advanced hepatocellular carcinoma. Biliary tract carcinoma are rare, accounting for about 3% of all digestive system malignancies. BTC are aggressive and were usually found in advanced stage, with a 5-year survival rate less than 5%. For advanced BTC, chemotherapy is the mainly systematic therapy recommended by current guidelines, targeted therapy and immunotherapy have shown efficacy in the exploration of the first-line and post-line of BTC. Anti-angiogenesis targeted drugs including lenvatinib are recommended for the first- or second-line treatment of advanced BTC.

Kidney injury is one of the common adverse reactions of anti-angiogenesis targeted drugs, among which proteinuria is one of the most common adverse reactions. Multiple key clinical studies have shown that the incidence of proteinuria associated with targeted therapy ranges from 10% to 51%, and the incidence of drug reduction or interruption due to proteinuria ranges from 0.9% to 17%.

Huaier is an extract from a medicinal fungus. The main effective component of Huai Qi Huang granule is Trametes Robiniophila Murr, which has been used in the treatment of chronic kidney disease for more than ten years. It was found that the effect of Huai Qi Huang granule alone or combined with RASI in the treatment of proteinuria was better than conventional treatment. The effective component of Huaier granule is also Trametes Robiniophila Murr, and its content is higher than that of Huai Qi Huang granule. Therefore, it is speculated that Huaier granule have a certain effect on anti-angiogenesis targeted therapy associated proteinuria in advanced hepatobiliary malignancies.

In this study, 1 research centers will participate. This study planned to enroll 53 participants. All the participants will be treated with Huaier granule. In this study, participants will be followed up for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years and older
2. Meeting the clinical diagnostic criteria of primary hepatobiliary malignancies, diagnosed as advanced hepatobiliary malignancies.
3. Receiving VEGFR-TKIs for advanced hepatobiliary malignancies.
4. Urinalysis indicates urine protein positive.
5. Urine protein level greater than 0.3 grams and less than 3.5 grams per 24 hours.
6. No Huaier granule were used within 1 month before enrollment.
7. Agree to use Huaier granule after enrollment.
8. Expected survival time not less than 6 months.
9. Volunteer to join the study and sign the informed consent form.

Exclusion Criteria:

1. Allergic to the components of Huaier granule, or avoid to use Huaier granule or use with caution.
2. Not able to take medication orally.
3. Must use or are using drugs that may affect proteinuria other than VEGFR-TKIs, including but not limited to bevacizumab, ACEI, glucocorticoids (more than 3 weeks), traditional Chinese medicine (refer to drug instructions).
4. Concomitant with other diseases that can lead to proteinuria, including but not limited to nephropathy, hypertension, urinary infections, systemic lupus erythematosus, multiple myeloma.
5. Pregnant or lactating women or women prepare for pregnancy.
6. Participating in clinical trials of other drugs that intend to treat proteinuria.
7. Refused to cooperate with follow-up.
8. Other reasons that the researcher considers unsuitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2025-09-16 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
The effective rate on proteinuria treatment after 8 weeks of Huaier granule | 8 weeks
  Proportion of subjects who achieved complete remission (CR) or partial remission (PR) or stable disease (SD) after 8 weeks treatment of Huaier granule.
  Perform a 24-hour urine collection for protein measurement, CR is defined as urine protein level≤0.3g/24h; PR is defined as urine protein level>0.3g/24h and<3.5g/24h, and decrease more than 30% from baseline; SD is defined as urine protein level >0.3g/24h and<3.5g/24h, and decrease less than or equal to 30% from baseline (or increase less than or equal to 20% from baseline); treatment failure is defined as at least two 24-hour urine protein tests show an increase of urine protein level of more than 20% from baseline or≥3.5 g/24h, or admission to renal replacement therapy or death.

SECONDARY OUTCOMES:
Mean value of 24-hour urinary protein level change from baseline to 8 weeks treatment of Huaier granule | 8 weeks
  Mean value of the difference between baseline 24h urine protein level and the 24h urine protein level after 8 weeks treatment of Huaier granule.
Mean value of 24-hour urinary protein level decrease rate from baseline to 8 weeks treatment of Huaier granule | 8 weeks
  Decrease rate: percentage of the difference between baseline 24h urine protein level and the 24h urine protein level after 8 weeks treatment of Huaier granule in baseline 24h urine protein level.
Incidence and severity of renal adverse events (AE) after 8 weeks treatment of Huaier granule | 8 weeks
Incidence and severity of serious renal adverse events (SAE) after 8 weeks treatment of Huaier granule | 8 weeks
Incidence and severity of renal adverse events (AE) after 16 weeks treatment of Huaier granule | 16 weeks
Incidence and severity of serious renal adverse events (SAE) after 16 weeks treatment of Huaier granule | 16 weeks

OTHER OUTCOMES:
Reduction rate of targeted drugs after 8 weeks treatment of Huaier granule | 8 weeks
  Proportion of subjects with VEGFR-TKIs drug reduction after 8 weeks treatment of Huaier granule.
Reduction rate of targeted drugs after 16 weeks treatment of Huaier granule | 16 weeks
  Proportion of subjects with VEGFR-TKIs drug reduction after 16 weeks treatment of Huaier granule.
Discontinuation rate of targeted drugs after 8 weeks treatment of Huaier granule | 8 weeks
  Proportion of subjects with VEGFR-TKIs drug discontinuation after 8 weeks treatment of Huaier granule.
4. Discontinuation rate of targeted drugs after 16 weeks treatment of Huaier granule | 16 weeks
  Proportion of subjects with VEGFR-TKIs drug discontinuation after 16 weeks treatment of Huaier granule.
ORR | 24 weeks
  Objective response rate: proportion of subjects who achieved complete remission (CR) or partial remission (PR) by primary tumor imaging evaluation.
DCR | 24 weeks
  Disease control rate: proportion of subjects who achieved complete remission (CR) or partial remission (PR) or stable disease (SD) by primary tumor imaging evaluation.
PFS | 24 weeks
  Progression free survival: time from the date when the subject first received targeted therapy he was receiving at the time of enrollment to the first observation of tumor progression or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Lu Wang, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No